CLINICAL TRIAL: NCT00693173
Title: Genital Drop Technique With Intensity-Modulated Radiation Therapy (IMRT) in Male Anal and Distal Rectal Cancer Patients: A Dosimetric Comparison
Brief Title: Radiation Dosimetry Study Comparing 2 Different Patient Setups in Anal/Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 07-049
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Anal Cancer
Keywords: anal; cancer; rectal; IMRT; genital; sparing; drop; technique
MeSH Terms: conditions — Anus Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study compares two patient setups (Standard Prone vs. Genital Drop Technique) with identical radiation treatment technique and parameters. After the two setups have been planned, the treating faculty reviews the setups and will choose the setup he feels that will give the patient improved dosimetry to the local regions and hopefully reduce toxicity and improve treatment tolerability.

DETAILED DESCRIPTION:
This is a study of two different setups when treating a patient with standard of care radiation doses. The study compares two patient setups (Standard Prone vs. Genital Drop Technique) with identical radiation treatment technique and parameters. After the two setups have been planned, the treating faculty reviews the setups and will choose the setup he feels that will give the patient improved dosimetry to the local regions and hopefully reduce toxicity and improve treatment tolerability.

Patients will not be randomized or stratified by demographic or disease risk assessment, but treatment will be tailored to stage specific current standards of care.

An extra (non standard of care) CT is required to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven anal cancer (squamous, basaloid, or cloacogenic carcinoma) or distal rectal cancer (adenocarcinoma variants) that traverse the dentate line and are eligible for definitive chemoradiation or preoperative radiation therapy, respectively.
* Any histological grade.
* Age: >18 years.
* Gender: Male patients with average external genitalia.
* Race: Any.
* Language: English speaking only.
* Performance status: Good (Karnofsky Performance Status of >60%). (ECOG 0-2).
* UTMB patients
* Stages: Early local disease to locoregionally advanced disease per the 2002 American Joint Committee on Cancer (AJCC) Staging System.
* Anal Cancer: Stages I-IIIB (see Section 11).
* Distal Rectal Cancers that pass the dentate line and into the anal canal only: Stages IIA-IIIC (see Section 11).

Exclusion Criteria

* Histological variants other than those listed above in 4.a.
* Patients with cystocele or abnormal scrotal edema will be excluded. (Although the Genital Drop Technique may specifically benefit this group of patients, however this study is to be performed with average patient anatomy).
* 2002 American Joint Committee on Cancer (AJCC) Staging System. (Anal Cancer: Stage IV.; Distal Rectal Cancer: Stage IV, and tumor 2-node 0-metastasis 0 (T1-T2N0M0) patients).
* Performance status: Poor (Karnofsky Performance Status of <60%). (ECOG 3-4).
* Non-English speaking patients.
* Prior pelvic radiation.
* Prior pelvic malignancy.
* Anal cancer/rectal cancer surgery, except for biopsy at study site.
* Patient's mental condition and social support is such that he can neither understand the nature of the protocol nor comply with its requirements.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male anal cancer and distal rectal cancer patients 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The Genital Drop Technique (IMRT-GD) decreased the radiation dose to the testicles scrotal skin and penile shaft compared to standard prone technique. | Day 1. Pretreatment analysis.
  The Genital Drop Technique (IMRT-GD) decreased the radiation dose to the testicles, scrotal skin and penile shaft compared to the standard conformal radiation therapy (CRT) and IMRT plans while preserving adequate planned target volume (PTV) dose coverage and homogeneity to the target organs in male anal cancer patients.

SECONDARY OUTCOMES:
Dosimetry comparison details. | Day 1. Pretreatment parameters.
  Testicular dose: Volume receiving 14 Gy was 90% with CRT, 64% with IMRT, and 3% with IMRT-GD.
  Testicular dose: Volume receiving 30 Gy was 54% with CRT, 26% with IMRT, and 0% with IMRT-GD.
  External genitalia dose: Volume receiving 14 Gy was 93% with CRT, 79% with IMRT, and 35% with IMRT-GD.
  External genitalia dose: Volume receiving 30 Gy was 75% with CRT, 31% with IMRT, and 12% with IMRT-GD.
  Planning Target Volume receiving full 54 Gy dose was 93% with CRT, 93% with IMRT, and 94% with IMRT-GD.

CONTACTS AND LOCATIONS:
Overall Officials: Grant R. Seeger, MD, Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (1):
- The University of Texas Medical Branch at Galveston, Galveston, Texas, United States